CLINICAL TRIAL: NCT02297932
Title: Physical Activity in Multiple Sclerosis (MS): A Novel Approach to Study Outcomes
Acronym: PHYSACTINMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Helen Genova, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 843-14
Record Dates: First submitted 2014-11-10; First posted 2014-11-21 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
Keywords: Exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength training (Experimental): The intervention will consist of a Home-based Resistant Training Intervention. Participants randomized to the home-based progressive resistance training (PRT) condition and will be provided with a training manual, an exercise log book, and resistance training equipment. The training manual will consist of a detailed description of the exercises to be performed and how to progress over 4-months. The exercise logbook will allow participants to provide a detailed recording of each training session. Home-based PRT equipment will consist of elastic bands (Thera-Band®, Hygenic Corporation, Akron, OH) and weighted vests.
  Interventions: Behavioral: Strength training
- Stretching (Active Comparator): Individuals in the comparator group will participate in a four month home-based stretching program developed by the National Multiple Sclerosis Society (NMSS). They will be provided text-based materials and asked to provide a weekly log book. In efforts to equate the attention received, individuals will come to KF at the same frequency as those receiving the PRT intervention and will also engage in the same number of sessions to assess their adherence to the program.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Strength training — Participants will engage in a home-based strength training program.
  Arms: Strength training
Behavioral: Stretching — Participants will engage in a home-based stretching training program
  Arms: Stretching

SUMMARY:
Physical activity and exercise interventions in multiple sclerosis (MS) have received great attention most recently and there exists several randomized clinical trials (RCTs) addressing the outcomes associated with such intervention. The majority of such interventions have primarily focused on directly influencing disease processes (e.g., inflammation, neurotrophic factors), the reduction of symptoms (e.g., fatigue, depression), improvement in physical functioning (e.g., gait, strength) or enhancing one's quality of life. To date, the evidence suggests that exercise intervention in MS holds anywhere from minimal to great promise depending on the outcome of interest. For some outcomes such as depression or cognition, findings are even less optimistic, being null, or inconsistent, at best. These inconsistent findings may be attributed to methodological issues such as use of subjective reports, lack of appropriate control group, poor compliance, and sample selection. The proposed investigation aims to address some of these issues by: (1) Obtaining objective measures of outcomes of interest (i.e., fatigue, cognition, and participation/activities of daily living [ADLs]) and; (2) assessing certain person-specific factors (e.g., personality) and intermediary factors that may be influenced by physical activity and indirectly result in improved outcomes (e.g., improvement in sleep and subsequent improvement in fatigue and/or cognition). Thus, the primary objective of the proposed investigation is to: (1) utilize innovative and objective measures of outcomes and; (2) obtain comprehensive assessment of intermediary variables (e.g., sleep) or person-specific characteristics (e.g., personality), which together may explain the inconsistent findings in the literature and has the following specific aims:

To achieve these goals, individuals will complete a comprehensive assessment of cognition, person-specific factors, intermediary factors, physical fitness, and functional magnetic resonance imaging (fMRI) prior to and following a home based exercise intervention.

DETAILED DESCRIPTION:
PROPOSAL NARRATIVE Specific Aims Specific Aim 1: Utilize innovative and objective measures/techniques (i.e., brain imaging, structured clinical interviews, performance based assessment of functional activity) to examine the effects of physical activity on fatigue, cognition, and participation/activities of daily living (ADLs).

Specific Aim 2: Obtain preliminary data to identify factors that may explain the inconsistencies in the literature pertaining to effects of physical activity on fatigue, cognition, and participation/ADLs. Specifically, intermediary factors may include sleep quality, depression, pain, and self-efficacy, which may be affected by the intervention and subsequently influence outcomes. Other potential factors that are independent of the intervention may include person-specific, baseline characteristics such as personality, trait anxiety, motivation, health beliefs and engagement in health-related behaviors, and certain demographics and disease variables (e.g., age).

Procedures. Subjects will be randomly assigned to either the strength training or stretching group based on an a priori randomization scheme. All participants will complete pre and post assessments consisting of subjective and objective measures of fatigue, cognition, & participation/ADLs (Per Specific Aim 1). Additionally baseline physical functioning measures will be included.

Fatigue Measures: Briefly, all imaging data for the study will be obtained using a 3.0 T Siemens Allegra scanner. The following anatomical images will be obtained: MPRAGE and localizer. fMRI will be performed during the performance of a cognitively fatiguing task (Modified SDMT [mSDMT]) during which the subject will be asked throughout the task to report on a scale of 0-100 how cognitively fatigued they feel "right now, at this moment." These ratings will then be used as an amplitude modulated regressor to determine where in the brain increased fatigue is associated with increased brain activity. Once this neural network is identified, we can compared the activation observed following the intervention.

Intervention. The intervention will consist of a Home-based Resistance Training Intervention. Participants randomized to the home-based progressive resistance training (PRT) condition and will be provided with a training manual, an exercise log book, and resistance training equipment. The training manual will consist of a detailed description of the exercises to be performed and how to progress over 6-months. The exercise logbook will allow participants to provide a detailed recording of each training session. Home-based PRT equipment will consist of elastic bands (Thera-Band®, Hygenic Corporation, Akron, OH) and weighted vests. This equipment has been used successfully in supervised and home-based PRT interventions which have improved strength, function, and health-related outcomes in clinical populations, particularly older adults. Participants will be involved in an initial training session at Kessler Foundation (KF) to learn how to perform the exercise program including demonstration and practice of exercise techniques, use of training equipment, and how to monitor and record training progress. Four follow-up visits to KF will occur throughout the 4-month program to provide participants with individualized feedback and training progressions. The home-based PRT program is based on the American College of Sports Medicine (ACSM) guidelines for prescription of resistance training, as well as previous PRT programs in persons with MS. This prescription is further consistent with recently developed evidence-based guidelines for physical activity for persons with MS. The prescription will consist of 3 weekly sessions of 1-3 sets, 8-12 repetitions of 10 exercises targeting lower body, upper body, and core muscle groups. The 10 exercises will include lunges, chair raises/squats, calf raises, knee flexion, knee extension, shoulder row, shoulder lateral raise, elbow flexion, elbow extension, and abdominal curls. The intensity of the training program will be prescribed based on the type or color of elastic band used and the amount of weight in the weighted vest, and is based on previous studies using these modalities.Five colors of elastic bands will be used which vary in level of resistance or difficulty (i.e., yellow < red < green < blue < black). Participants will begin with the yellow band and progress following the described color band progression. The amount of weight added to the weighted vest will be determined as a percent of each individual's body weight. The initial weight in the vest will be set as 0.5% of body weight. Vest weight progression will occur by adding 0.5 to 1.5% of body weight every 2 weeks for the first 12 weeks of the program. During the second half of the program, vest weight progression will occur by adding 0.05 to 1.0% of body weight every 2 weeks. At each follow-up training session, body weight will be re-assessed to ensure accurate training progression. Other progressions throughout the program will include increasing the number of sets and repetitions, and increasing the level of difficulty of the exercises (e.g., changing exercise position from sitting to standing). Individualized feedback and progress with the program will be provided during one-on-one phone chat sessions. This will provide participants with the opportunity to modify and adapt their goals as they progress through the program with the ultimate goal of developing the skills necessary to independently monitor and change their behavior. The behavioral content will be delivered through text-based materials and one-on-one phone chat sessions with a member of the research team not involved in outcome assessments. Text-based materials will be provided at the initial training session including the training manual, exercise log book, and information on self-monitoring and setting goals for the PRT program.

Comparison Group. Individuals in the stretching condition will participate in a four month home-based stretching program developed by the National Multiple Sclerosis Society (NMSS). They will be provided text-based materials and asked to provide a weekly log book. In efforts to equate the attention received, individuals will come to KF at the same frequency as those receiving the PRT intervention and will also engage in the same number of chat sessions to assess their adherence to the program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis (MS).
* Ability to read and speak English fluently.
* Ability to walk independently without the use of any assistive devices (e.g. cane, walker, or wheelchair).

Exclusion Criteria:

* Left handedness
* Presence of a clip to repair a cerebral aneurysm (broken blood vessel in the head), cardiac pace-maker, cochlear implants (internal hearing aids) or metal fragments or pieces in eyes or any other part of body.
* Non MRI compatible metal in any part of body.
* Physician's instruction that it is medically unsafe for subject to receive regular MRI as part of their medical care.
* Engagement in the professions of painting or welding or other occupation that precludes an individual from getting a regular MRI.
* Proneness to claustrophobia (fear of enclosed spaces), to my knowledge.
* History of schizophrenia or bipolar disorder.
* Pregnancy
* History of stroke, brain Injury or neurological disease other than MS.
* Evidence of a flare up of MS symptoms within the past month.
* Administration of the following in last month: steroids, benzodiazepines, neuroleptics or opiates, as determined by the study doctor.
* History of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of serious depression requiring treatment with medication,, Schizophrenia, Bipolar Disorder I or II.
* Significant alcohol or drug abuse history

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fatigue after 4-month exercise intervention (Questionnaires and fMRI) | Baseline and post-4 month intervention
  Subjective: Questionnaires; Objective: fMRI during performance of a cognitively fatiguing task
Change from baseline in cognition after 4-month exercise intervention (Questionnaires and neuropsychological testing) | Baseline and post-4 month intervention
  Subjective: Questionnaire; Objective: Standardized neuropsychological testing
Change from baseline in participation in activities of daily living (ADLs) after 4-month exercise intervention (Questionnaire; The Neistadt and Crepeau Activities of Daily Living test; Timed Instrumental Activities of Daily Living (TIADL) test | Baseline and post-4 month intervention
  Subjective: Questionnaire; Objective : The Neistadt and Crepeau Activities of Daily Living test; Timed Instrumental Activities of Daily Living (TIADL) test

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Weiner, Study Director — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States